CLINICAL TRIAL: NCT03681119
Title: The Hospice Advanced Dementia Symptom Management and Quality of Life Trial (HAS-QOL)
Brief Title: The Hospice Advanced Dementia Symptom Management and Quality of Life Trial
Acronym: HAS-QOL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 18-01265
Record Dates: First submitted 2018-09-20; First posted 2018-09-21 (Actual); Results first posted 2020-07-23 (Actual); Last update posted 2020-08-13 (Actual); Status verified 2020-08

CONDITIONS: Dementia
MeSH Terms: conditions — Dementia | interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Advanced Demential Patients (Experimental)
  Interventions: Behavioral: Dementia symptom management at home hospice edition
- Hospice IDT Members (Experimental)
  Interventions: Behavioral: Education and Training

INTERVENTIONS:
Behavioral: Dementia symptom management at home hospice edition — Quality assurance performance improvement program
  Arms: Advanced Demential Patients
Behavioral: Education and Training — Education and training
  Arms: Hospice IDT Members

SUMMARY:
Alzheimer's Disease and Related Disorders (dementia) are a group of serious life limiting illness that cause significant challenges to our public health system, with significant illness burden for both the person with dementia and the caregiver. At the end of life, over 230,000 persons with dementia annually are cared for in hospice, yet hospice agencies are ill prepared to care for this population and often resort to inappropriate pharmacologic measures such as antipsychotics that reduce quality of life rather than improve it. This study will therefore through its two phases refine and then implement, using a pragmatic stepped wedge trial design, the Dementia Symptom Management at Home Program Hospice Edition, with the goal improving quality of care for the person with dementia and their caregiver, reducing antipsychotic use, and increasing bereaved caregiver satisfaction in the hospice setting.

ELIGIBILITY:
Inclusion Criteria:

* Must have dementia as primary diagnosis for admission to hospice
* Must be newly admitted to a participating hospice
* Must be 50 years or older

Clinicians:

* Must be a skilled clinician or home health aide who provides care through an eligible home health agency
* Must be 18 years or older

Exclusion Criteria:

Persons with Dementia:

* None

Clinicians:

* None

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2019-02-11 (Actual); Primary Completion 2019-06-12 (Actual); Study Completion 2019-06-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Abraham Brody, PhD, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification.
Supporting Information: Study Protocol
Time Frame: Beginning 3 months and ending 5 years following article publication.
Access Criteria: Researchers who provide a methodologically sound proposal.

REFERENCES:
- [Derived] Lin SY, Schneider CE, Bristol AA, Clancy M, Sprague SA, Aldridge M, Cortes T, Goldfeld KS, Kutner JS, Mitchell SL, Shega JW, Wu B, Zhu CW, Brody AA. Findings of Sequential Pilot Trials of Aliviado Dementia Care to Inform an Embedded Pragmatic Clinical Trial. Gerontologist. 2022 Feb 9;62(2):304-314. doi: 10.1093/geront/gnaa220. PMID 33377138
- [Derived] Schneider CE, Bristol A, Ford A, Lin SY, Palmieri J, Meier MR, Brody AA; HAS-QOL Trial Investigators. The Impact of Aliviado Dementia Care-Hospice Edition Training Program on Hospice Staff's Dementia Symptom Knowledge. J Pain Symptom Manage. 2020 Aug;60(2):e7-e13. doi: 10.1016/j.jpainsymman.2020.05.010. Epub 2020 May 15. PMID 32416231

RESULTS

PARTICIPANT FLOW:
Groups:
- Hospice IDT Members: Hospice Interdisciplinary Team (IDT)
Period: Overall Study
Arm/Group | Hospice IDT Members | Advanced Demential Patients
Started | 72 | 11
Completed | 66 | 11
Not Completed | 6 | 0
Not completed — No specific reason | 4 | 0
Not completed — Sickness | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Hospice IDT MembersHospice Clinicians (RNs, Social Workers, Ch: Hospice Clinicians (RNs, Social Workers, Chaplains) who are given training
- Total: Total of all reporting groups
Arm/Group | Hospice IDT MembersHospice Clinicians (RNs, Social Workers, Ch | Advanced Demential Patients | Total
Number analyzed (Participants) | 72 | 11 | 83
Age, Continuous [Mean (Full Range); unit: years] | 50.7 [29 to 74] | 86 [56 to 94] | 68.4 [29 to 94]
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Sex: Female | 57 | 11 | 68
  Sex: Male | 9 | 0 | 9
  Sex: Unknown or not reported | 6 | 0 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 0 | 5
  Not Hispanic or Latino | 67 | 11 | 78
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 6 | 1 | 7
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 19 | 0 | 19
  White | 23 | 10 | 33
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 22 | 0 | 22

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Hospice IDT Members Who Complete Required Education and Training
Description: Percentage of Hospice IDT Members who Complete Required Education and Training
Time Frame: 2 Months
Measure: Number; unit: percentage of participants
Groups:
- Hospice IDT Members: Hospice Clinicians (RNs, Social Workers, Chaplains) who are given training
Arm/Group | Hospice IDT Members
Number analyzed (Participants) | 72
percentage of participants | 92

ADVERSE EVENTS:
Time Frame: 1 month
Description: All qualifying adverse events were pulled from all eligible patients' electronic health records. Adverse events were only reported on the Advanced Dementia Patients arm.
Arm/Group | Advanced Demential Patients
All-Cause Mortality (participants affected / at risk) | 5/11
Serious Adverse Events (participants affected / at risk) | 5/11
Other Adverse Events (participants affected / at risk) | 0/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Advanced Demential Patients (N=11)
Death (Nervous system disorders) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-28): https://cdn.clinicaltrials.gov/large-docs/19/NCT03681119/Prot_SAP_000.pdf